CLINICAL TRIAL: NCT01910532
Title: The Evaluation of Clevidipine in Patients Requiring ICP Monitoring and IV Antihypertensive Therapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor discontinued the research
Sponsor: Mario Ammirati (Other)
Responsible Party: Sponsor-Investigator, Mario Ammirati, Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009H0336
Record Dates: First submitted 2011-12-19; First posted 2013-07-29 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clevidipine (Experimental): Using Clevidipine for the treatment of acute hypertension defined SBP > 160 mmHg in patients who require an Intracranial Pressure Monitoring Device
  Interventions: Drug: Clevidipine

INTERVENTIONS:
Drug: Clevidipine — Clevidipine for the treatment of acute hypertension defined SBP > 160 mmHg in patients who require an Intracranial Pressure Monitoring Device

SUMMARY:
This is a single-arm, open label safety and dose titration study evaluating the use of Clevidipine to rapidly control elevated blood pressure in patients who have an Intracranial Pressure Monitoring device.

DETAILED DESCRIPTION:
This is a single-arm, open label safety and dose titration study evaluating the use of Clevidipine to rapidly control elevated blood pressure in patients who have an Intracranial Pressure Monitoring device.

All patients in which ICP monitoring is carried out need to maintain Cerebral Perfusion Pressure (CPP) within a tight range (typically, 70-90 mmHg) in order to avoid secondary brain injuries related to either too high or too low CPP. In this context there are clear benefits associated with a medication that is able to control hypertensive situations quickly and that lends itself to easy and reliable modulation.

Clinical studies have demonstrated that Clevidipine is an effective antihypertensive agent with a rapid onset and offset of action, and a favorable safety profile. Clevidipine has a predictable dose-response profile and is readily titrated to achieve individualized pharmacodynamic effects.

The investigators reasoned that Clevidipine could be an effective anti-hypertensive agent in this cohort of patients in which there is a need for rapid and precise blood pressure control. It is further hypothesized that improved blood pressure control in this patient population may result in the reduction in the severity of their neurological impairment.

The question to be answered is as follows: Is Clevidipine highly effective in achieving and maintaining Blood Pressure control in patients with hypertension (Systolic Blood Pressure > 160 mm Hg) and who require an Intracranial Pressure Monitoring Device?

Clevidipine will be highly effective in achieving and maintaining Blood Pressure control in patients with hypertension and who require an Intracranial Pressure Monitoring Device.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years or older
2. Written informed consent from the patient or their legal representative family member before initiation of any study-related procedures
3. Patients who clinically require Intracranial Pressure Monitoring device
4. Patients who have baseline systolic blood pressure (SBP) (immediately prior to initiation of Clevidipine) > 160 mmHg measured using an arterial line
5. Patients who required IV antihypertensive therapy to achieve SBP ≤ 160 mm Hg

Exclusion Criteria:

1. Patients who are prisoners
2. Patients who received an oral antihypertensive medication within 2 hours prior to initiation of Clevidipine
3. Patients who received any other IV antihypertensive medication within 2 hours prior to initiation of Clevidipine
4. Patients who have fixed dilated pupils and/or absence of gag and oculo-cephalic brain stem reflexes
5. Patients with a history of allergy or intolerance to calcium channel blockers
6. Patients with a history of allergy to soybean oil or egg lecithin
7. Patients who have participated or are currently participating in a clinical trial of an investigational drug within 30 days prior to enrollment
8. Patients who have acute myocardial infarction (AIM) on presentation
9. Patients who have known or suspected aortic dissection
10. Females who are pregnant or are breastfeeding
11. Patients with a history of liver failure, cirrhosis or pancreatitis
12. Patients with a prior directive against advanced life support
13. Patients with a history of impaired lipid metabolism
14. Patients with a history of severe aortic stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Time to achieve target Systolic Blood Pressure within 30 minutes of start of Celevidipine infusion | Up to 1 year
  To evaluate the efficacy of Clevidipine for the treatment of acute hypertension during the first 30 minutes after initiation of the intravenous infusion in patients who require an Intracranial Pressure Monitoring Device

SECONDARY OUTCOMES:
Percentage of patients who reach target Systolic Blood Pressure within 30 minutes of start of Clevidipine infusion | Up to 1 year
  To evaluate the efficacy of Clevidipine to maintain Systolic Blood Pressure (SBP) within the target range after the first 30 minutes of an initial infusion and up to 3 hours in patients who required an Intracranial Pressure Monitoring
Percentage of patients in who the Systolic Blood Pressure is maintained within the target range for up to 3 hours after the first 30 minutes of the start of Clevidipine infusion | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mario Ammirati, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States